CLINICAL TRIAL: NCT05264090
Title: Seven-day Ambulatory Blood Pressure Monitoring and CAVI in the Prevention of Cardiovascular Diseases
Brief Title: Possibilities of Interpreting the Night-to-Day Ratio Specified by 24-hour Blood Pressure Monitoring
Acronym: ABPM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Anne's University Hospital Brno, Czech Republic (Other)
Collaborators: Masaryk University (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 24H7D_ABPM
Record Dates: First submitted 2022-02-09; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Cardiovascular Diseases
Keywords: ambulatory blood pressure monitoring; hypertension; night-to-day ratio; exercise
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Motor Activity

STUDY DESIGN:
Intervention Model Description: Monocenter, non-randomized, controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Placebo Comparator): Healthy volunteers without exercise
  Interventions: Other: Ambulatory blood pressure monitoring
- Group 2 (Sham Comparator): Healthy exercise-training volunteers
  Interventions: Other: Ambulatory blood pressure monitoring; Other: Combined aerobic-resistance exercise
- Group 3 (Active Comparator): Patients with ischemic coronary artery disease without exercise
  Interventions: Other: Ambulatory blood pressure monitoring
- Group 4 (Experimental): Patients with ischemic coronary artery disease following cardiovascular rehabilitation
  Interventions: Other: Ambulatory blood pressure monitoring; Other: The cardiovascular exercise

INTERVENTIONS:
Other: Ambulatory blood pressure monitoring — The ambulatory monitoring (7-day ABPM) was performed with ambulatory blood pressure monitoring devices TM-2430 (A&D; Tokyo, Japan) based on both the cuff-oscillometric and Korotkoff sound method. The cuff was placed on the non-dominant arm according to the same rules applying to casual auscultation measurement. The monitoring device with a weight of 250 g was worn by the monitored subjects in a waist-fixed case continuously for 7 days except for times involving personal hygiene. During every automatic measurement, the arm was resting and hung along the body. The device automatically recorded all the regular measurements for seven days, between 6:00 a.m. and 10:00 p.m. every 30 minutes and between 10:00 p.m. and 6:00 a.m. every 60 minutes. Such short intervals are necessary to obtain a sufficient number of representative measurements.
Other: Combined aerobic-resistance exercise — Combined aerobic-resistance exercise (group 2) was scheduled twice weekly in the form of 60-minute workouts with a load intensity at the level of sub-maximum heart frequency (75-85% SFmax). The minimum time span between the workouts was 24 hours. The workout consisted of a 10-minute warm-up, 25 minutes of aerobic exercise (spinning bicycle or bicycle ergometer), 15 minutes of resistance exercise on gym machines (bench press, leg extension and pull down) with 40-50% 1-RM (one repetition maximum) intensity (3 series of 10 exercises), and a 10-minute cool-down (stretching of the main muscle groups).
  Arms: Group 2
Other: The cardiovascular exercise — The cardiovascular exercise (group 4) took the form of sixty-minute workouts scheduled two to three times weekly. The nature of the workouts was similar, combined aerobic-resistance exercise (a 10-minute warm-up, aerobic endurance on bicycle ergo meter for 25 minutes, resistance exercise on multifunctional gym machines for 15 minutes, and a 10-minute cool-down). The workout intensity was set at the level of the first ventilation threshold (VAT-1), corresponding to the following workout parameters: load (W) and heart rate (HR).19,20 The resistance exercise intensity was specified by the 1-RM (one repetition maximum) method. The maximum load lifted across the full range of motion for every exercise was used as the benchmark for the workload intensity specification, corresponding to 30 - 60% 1-RM.
  Arms: Group 4

SUMMARY:
Specify the risk rate of incorrect patient classification based on night-to-day ratio specification from singular 24-h ABPM in comparison to the results of 7-day ABPM monitoring

DETAILED DESCRIPTION:
The subjects in the study are divided into 4 groups:

group 1 (40 healthy men and women without exercise); group 2 (40 healthy exercise-training men and women); group 3 (40 patients with ischemic coronary artery disease without exercise); and group 4 (51 patients with ischemic coronary artery disease following cardiovascular rehabilitation).

The subject of the evaluation is the percentage rate of incorrect subject classification (dipper, non-dipper, extreme dipper, and risers) based on the mean blood pressure values for 7 days and from seven independent 24-hour cycles (the mean value mode).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (without any disease, including the cardiovascular ones, and without any kind of treatment)
* Patients with chronic ischemic coronary artery disease
* Patients treated with ACE inhibitors, beta-blockers or statins.
* To visit routinely in the health centres where the study is carried out

Exclusion Criteria:

* Age under 18 years,
* Pregnant, or breast-feeding,
* Patients on dialysis or being followed by nephrology,
* Severe physical or cognitive limitations,
* Intolerance to the method of measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
The risk rate of incorrect patient classification based on night-to-day ratio specification from singular 24-h ABPM in comparison to the results of 7-day ABPM monitoring. | 1 - 7 days
  Primary outcome was to specify the risk rate of incorrect patient classification based on night-to-day ratio specification from singular 24-h ABPM in comparison to the results of 7-day ABPM monitoring.
  The percentage of blood pressure drop at night expressed by night-to-day ratio (dippers, non-dippers, extreme dippers, reverse dippers) can be specified much more accurately on the basis of 7-day ABPM values. ABPM restricted to 24 h, as currently practiced, does not yield a sufficiently reliable estimate of the night-to-day ratio for a classification in terms of dipping. Extending monitoring to 7 days accounts for the large day-to-day variability in the night-to-day ratio, and may yield a more reliable diagnosis of blood pressure variability.

SECONDARY OUTCOMES:
Optimalization of the blood pressure diagnostic through comparing of 24 hours and 7 days monitoring. | 1 - 7 days
  On the basis of the obtained results, the following procedure can be recommended for clinical practice. If the standard 24-hour monitoring is used, then obtain at least 3 mutually independent 24-hour cycle data for every examined individual. If at least two of them result in the same night-to-day ratio and the third night-to-day ratio is only slightly different, the thus obtained index can be considered trustworthy. Otherwise, the correct night-to-day ratio can only be obtained by 7-day ABPM and, in addition, the resulting night-to-day ratio calculated from the mean values obtained in the course of the 7 days must be compared to the result modes obtained for the individual monitoring days.
  The magnitude of the difference between the evaluation of 24-hour and 7-days blood pressure records was not dependent on the gender, age, health, or cardiovascular disease or physical activity of monitored individuals.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Anne´s University Hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No